CLINICAL TRIAL: NCT02938247
Title: Prospective Tolerance and Compliance Study With a High Caloric, High Protein Oral Nutritional Supplement in Nursing Home Residents - Scheduled Intake
Brief Title: Tolerance and Compliance of a High Caloric, High Protein Oral Nutritional Supplement - Scheduled Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: F3kc-002-CNI
Record Dates: First submitted 2016-09-12; First posted 2016-10-19 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Malnutrition
Keywords: Malnutrition; Geriatric subjects; Nursing home
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm study (Experimental): High caloric, high protein ONS, three portions daily, total dose of 400 kcal/day for 7 consecutive days, oral administration
  Interventions: Dietary Supplement: High caloric, high protein ONS

INTERVENTIONS:
Dietary Supplement: High caloric, high protein ONS

SUMMARY:
The aim of the study is to assess gastro-intestinal tolerance, palatability, compliance, and use of a high caloric, high protein oral nutritional supplement (ONS) in elderly people

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male/female
2. Age: 65 years or older
3. Body-mass index (BMI): ≥ 16.0 kg/m² and ≤ 30.0 kg/m²
4. Subjects with an indication for ONS of approx. 400 kcal per day for at least 7 days
5. Written informed consent

Exclusion Criteria:

1. Existing gastrointestinal diseases or pathological findings, which do not allow enteral nutrition
2. Subjects with galactosaemia or similar metabolic disorders
3. Subjects with severely impaired gastrointestinal function or complete failure
4. Subjects with insulin-requiring diabetes
5. Subjects with acute diarrhoea (defined as ≥ 3 loose or watery stools per day)
6. Subjects reporting frequent occurrence of migraine attacks
7. Subjects with acute or (current) chronic diseases, which might lead to impaired gustatory sense (e.g. sinusitis, anosmia)
8. Existing mouth abnormalities, which cause impaired gustatory sense
9. Subjects who report impaired gustatory sense (e.g. due to intake of concomitant medication)
10. Subjects passing through chemotherapy (last cycle < 2 months ago)
11. Known allergic reactions or intolerance to any ingredient used or to constituents of the ONS
12. Subjects with severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical study by the investigator
13. Consumption of any additional ONS, enteral nutrition via tube or parenteral nutrition
14. Subjects with need of a special diet contradicting the intake of the ONS
15. History of relevant central nervous system (CNS) and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
16. Subjects with dysphagia or with high aspiration risk
17. Enrolment in another clinical study
18. Administration of any investigational medicinal product during the last month prior to individual enrolment of the subject
19. Subjects who are not able to self-report GI-problems and compliance
20. Subjects who report a general dislike of the ONS flavour
21. Subjects for whom a hospitalisation for rehabilitation or surgery during the study is planned
22. Subjects suspected or known not to follow instructions
23. Subjects unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Gastro-intestinal (GI) tolerance assessed by investigator (physical examination / presence of GI symptoms) | At screening examination (study days -3 to -1)
  The presence of the following GI symptoms will be documented: diarrhoea, constipation, bloating, distension, nausea, vomiting, burping, regurgitation, flatulence, abdominal discomfort, abdominal pain
Gastro-intestinal (GI) tolerance assessed by investigator (physical examination / presence of GI symptoms) | At end of study (study day 8)
  The presence of the following GI symptoms will be documented: diarrhoea, constipation, bloating, distension, nausea, vomiting, burping, regurgitation, flatulence, abdominal discomfort, abdominal pain
Gastro-intestinal (GI) tolerance assessed by subject (presence of GI symptoms assessed by subject's questionnaire) | At study days 1-8
  The presence of the following GI symptoms will be documented: diarrhoea, constipation, bloating, distension, nausea, vomiting, burping, regurgitation, flatulence, abdominal discomfort, abdominal pain

SECONDARY OUTCOMES:
Palatability of ONS (assessed by subject's questionnaire by using a 5-point hedonic-scale) | At study days 1 and 7
  Assessment of palatability (using a 5-point hedonic-scale) regarding appearance, smell, taste, sweetness, mouthfeel and product in general
Compliance assessed by comparison of ONS amount prescribed vs. actual intake (in mL) | At study days 1-7
Compliance assessed by comparison of ONS amount prescribed vs. actual intake (in %) | At study days 1-7
Compliance assessed by percentage of subjects who reached ≥ 75% of prescribed dose of ONS | At study days 1-7
Use of ONS assessed by consumption | At study days 1-7
  Confirmation of consumption under supervision of study team
Use of ONS assessed by presentation | At study days 1-7
  Confirmation of serving temperature
Reasons for non-compliance of ONS at a specific time of the day or on a specific day or for early termination (provided by subject by open question) | At study days 1-7
Reasons for non-use of ONS at a specific time of the day or on a specific day or for early termination (provided by subject by open question) | At study days 1-7

OTHER OUTCOMES:
Adverse Events | At study days 1-8

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius Koch, MD, Principal Investigator — SocraTec R&D GmbH, Clinical Pharmacology Unit
Locations (1):
- SocraTec R&D GmbH, Clinical Pharmacology Unit, Erfurt, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No